CLINICAL TRIAL: NCT05442190
Title: Phase 2 Study Evaluating SGX302 (Synthetic Hypericin) in the Treatment of Mild-to-Moderate Psoriasis
Brief Title: Topical SGX302 for Mild-to-Moderate Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HPN-PSR-01
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis; Plaque Psoriasis; Psoriasis Vulgaris
Keywords: Hypericin
MeSH Terms: conditions — Psoriasis | interventions — hypericin

STUDY DESIGN:
Intervention Model Description: This is a 2 part study. All protocol procedures, timing for schedule of events and assessments are identical for Parts A and B. In Part A, 10-15 patients will be assigned open-label SGX302 (ointment or gel). Once the tolerability and response to SGX302 has been established, Part B of the protocol will commence. In Part B, approximately 32 patients will be randomized to double-blind treatment groups at a ratio 1:1 of active drug to a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SGX302 Ointment (0.25 % Hypericin) (Experimental): SGX302 (0.25 % hypericin) ointment will be applied to lesions and treated with visible light 24±6 hours later starting at 5 J/cm^2. Drug application/light session will be done twice a week (at least 2 calendar days apart) for 18 weeks.
  Interventions: Drug: Hypericin
- Placebo (Ointment without Hypericin) (Placebo Comparator): Placebo ointment will be applied to lesions and treated with visible light 24±6 hours later starting at 5 J/cm^2. Drug application/light session will be done twice a week (at least 2 calendar days apart) for 18 weeks.
  Interventions: Drug: Placebo
- SGX302 Gel (0.25 % hypericin) (Experimental): SGX302 (0.25 % hypericin) gelt will be applied to lesions and treated with visible light 24±6 hours later starting at 5 J/cm^2. Drug application/light session will be done twice a week (at least 2 calendar days apart) for 18 weeks.
  Interventions: Drug: Hypericin

INTERVENTIONS:
Drug: Hypericin — SGX302 is synthetic hypericin formulated as a 0.25% hypericin ointment or gel.
  Other Names: SGX302
  Arms: SGX302 Gel (0.25 % hypericin); SGX302 Ointment (0.25 % Hypericin)
Drug: Placebo — Placebo ointment is identical to SGX302 ointment (color matched) but it does not contain hypericin.
  Arms: Placebo (Ointment without Hypericin)

SUMMARY:
To evaluate SGX302 (topical hypericin ointment and gel) with visible light in an initial 18-week treatment course for improving lesions in patients with mild-to-moderate psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of plaque psoriasis (psoriasis vulgaris) of at least 6-months duration that involves the body (trunk and/or limbs) that is amenable to topical treatment and opaque coverage after application.
* Have a static Investigator Global Assessment (IGA)/Psoriasis Area and Severity Index (PASI) of disease severity of mild or moderate on the body (trunk and/or limbs).
* Have lesions involving 2-30% of the body (trunk and/or limbs). For subjects with scalp psoriasis included in the treatment area, the total treatment area on body and scalp must not exceed 30%.

Exclusion Criteria:

* Use of topical anti psoriatic therapy within one week prior to the beginning of the study and willing to not use other psoriasis treatments for 4 weeks following completion of the treatment portion of the study.
* Received systemic biologic therapy to treat psoriasis within 12 weeks prior to the beginning of the study.
* Received systemic psoriasis therapy within 4 weeks prior to the beginning of the study.
* Received phototherapy (including laser) or photodynamic (light activated drug) therapy within 4 weeks prior to the beginning of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Number of patients that achieve a 0 or 1 score using the 5-point Investigator's Global Assessment scale | 18 weeks
  The percentage of patients in each treatment group that achieve a 0 or 1 score (Clear or Almost Clear) evaluation using the 5-point Investigator's Global Assessment (IGA) scale.
  The 5-point IGA scale:
  * Score 0: Clear - No signs of psoriasis; post-inflammatory hyperpigmentation may be present
  * Score 1: Almost Clear - No thickening; normal to pink coloration; no to minimal focal scaling
  * Score 2: Mild - Just detectable to mild thickening; pink to light red coloration; predominantly fine scaling
  * Score 3: Moderate - Clear distinguishable to moderate thickening; dull to bright red; moderate scaling
  * Score 4: Severe - Severe thickening with hard edges; bright to deep red coloration; severe/coarse scaling covering almost all lesions

SECONDARY OUTCOMES:
Number of patients achieving a ≥75% improvement in Psoriasis Area and Severity Index | 18 weeks
  The percentage of patients in each treatment group that achieve a ≥75% improvement in Psoriasis Area and Severity Index (PASI 75).
  PASI is a combined assessment of lesion severity and affected area into a single score. The body is divided into 4 areas for scoring: head, arms, trunk and legs. Each area is scored by itself and scores are combined for a final PASI. For each area, scores of erythema, thickness and scale are scored on a scale of 0 (clear) to 4 (maximum). For each area, percent of skin involved is estimated: 0 = 0%, 1= 0 to ≤10%, 2 = 10 to <30%, 3 = 30 to <50%, 4 = 50 to <70%, 5 = 70 to ≤90%, 6 = 90 to100%. Final PASI = (sum of severity parameters for each area)*(area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4)).
Number of patients achieving a ≥90% improvement in Psoriasis Area and Severity Index | 18 weeks
  The percentage of patients in each treatment group that achieve a ≥90% improvement in Psoriasis Area and Severity Index (PASI 90).
  The calculation of PASI was previously described.
Number of patients achieving a 100% improvement in Psoriasis Area and Severity Index | 18 weeks
  The percentage of patients in each treatment group that achieve a 100% improvement in Psoriasis Area and Severity Index (PASI 100).
  The calculation of PASI was previously described.

CONTACTS AND LOCATIONS:
Locations (1):
- Therapeutics Clinical Research, San Diego, California, United States